CLINICAL TRIAL: NCT02676778
Title: A Phase 2 Study of E7777 in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma and Cutaneous T-cell Lymphoma
Brief Title: Study of E7777 in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma and Cutaneous T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7777-J081-205
Record Dates: First submitted 2016-02-04; First posted 2016-02-08 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Peripheral T-cell Lymphoma; Cutaneous T-cell Lymphoma
Keywords: Peripheral T-cell lymphoma; Cutaneous T-cell lymphoma; E7777; Phase 2
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous | interventions — E7777 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E7777 (Experimental): Participants with relapsed or refractory peripheral T-cell lymphoma (PTCL) and cutaneous T-cell lymphoma (CTCL) will receive 9 μg/kg/day of E7777, administered by intravenous drip infusion in 60 minutes (± 10 min) for Days 1 through 5 of each cycle in maximum of 8 cycles. Every cycle consists of 3 weeks.
  Interventions: Drug: E7777

INTERVENTIONS:
Drug: E7777

SUMMARY:
The purpose of this study is to evaluate the objective response rate (ORR) of E7777 in participants with relapsed or refractory peripheral T-cell lymphoma (PTCL) and cutaneous T-cell lymphoma (CTCL).

DETAILED DESCRIPTION:
This is a multicenter, single-arm, open label, Phase 2 to evaluate efficacy, safety, pharmacokinetics and immunogenicity of E7777 in participants with relapsed or refractory PTCL and CTCL.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have histological diagnosis as peripheral T-cell lymphoma (PTCL) and cutaneous T-cell lymphoma (CTCL).
2. Participant who have measurable disease.
3. Participant who had previous systemic chemotherapy.
4. Participant who had disease progression (PD) or did not have response (complete response (CR) or partial response (PR)) in systemic chemotherapy, or relapsed or progressed after systemic chemotherapy.
5. Participant with Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
6. Participant with adequate renal, liver and bone marrow function.
7. Male and female participants ≥20 years of age at the time of informed consent.
8. Participants who have provided written consent to participate in the study.

Exclusion Criteria:

1. Participant with serious complications or histories.
2. Participant with history of hypersensitivity to protein therapeutics.
3. Participant who is positive for Human immunodeficiency virus (HIV) antibody, Hepatitis C virus (HCV) antibody, or Hepatitis B Surface (HBs) antigen.
4. Participant with malignancy of activity other than PTCL or CTCL within 36 months before informed consent.
5. Women of childbearing potential or man of impregnate potential who don't agree to use a medically effective method for contraception.
6. Woman who is pregnant or lactating.
7. Participant with allogeneic stem cell transplantation.
8. Participant who were decided as inappropriate to participate in the study by the investigator or sub-investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- Japan (20):
  - Eisai Trial Site #1, Nagoya, Aichi-ken
  - Eisai Trial Site #2, Nagoya, Aichi-ken
  - Eisai Trial Site #1, Kashiwa, Chiba
  - Eisai Trial Site #1, Ōta, Gunma
  - Eisai Trial Site #1, Kobe, Hyōgo
  - Eisai Trial Site #1, Tsukuba, Ibaraki
  - Eisai Trial Site #1, Isehara, Kanagawa
  - Eisai Trial Site #1, Sendai, Miyagi
  - Eisai Trial Site #1, Kurashiki, Okayama-ken
  - Eisai Trial Site #1, Suita, Osaka
  - Eisai Trial Site #2, Suita, Osaka
  - Eisai Trial Site #1, Hamamatsu, Shizuoka
  - Eisai Trial Site #1, Yamagata, Tamagata
  - Eisai Trial Site #1, Bunkyo-ku, Tokyo
  - Eisai Trial Site #1, Chuo-ku, Tokyo
  - Eisai Trial Site #1, Koto-ku, Tokyo
  - Eisai Trial Site #1, Fukuoka
  - Eisai Trial Site #1, Kagoshima
  - Eisai Trial Site #1, Kyoto
  - Eisai Trial Site #1, Okayama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 20 investigative sites in Japan from 28 March 2016 to 26 April 2019.
Pre-assignment Details: A total of 45 participants were enrolled (obtained informed consent and screened), of these 8 were screen failures and 37 were treated.
Groups:
- PTCL: E7777 9 mcg/kg/Day: Participants with relapsed or refractory peripheral T-cell lymphoma (PTCL) received E7777 9 microgram per kilogram per day (mcg/kg/day) as intravenous infusion, once daily from Day 1 through Day 5 in each treatment cycle until discontinuation or Cycle 8 (each Cycle length equal to [=] 3 weeks).
- CTCL: E7777 9 mcg/kg/Day: Participants with cutaneous T-cell lymphoma (CTCL) received E7777 9 mcg/kg/day as intravenous infusion, once daily from Day 1 through Day 5 in each treatment cycle until discontinuation or Cycle 8 (each Cycle length = 3 weeks).
- Other: E7777 9 mcg/kg/Day: Participant with extranodal natural killer (NK)/T-cell lymphoma received E7777 9 mcg/kg/day as intravenous infusion, once daily from Day 1 through Day 5 in each treatment cycle until discontinuation or Cycle 8 (each Cycle length = 3 weeks).
Period: Overall Study
Arm/Group | PTCL: E7777 9 mcg/kg/Day | CTCL: E7777 9 mcg/kg/Day | Other: E7777 9 mcg/kg/Day
Started | 17 | 19 | 1
Completed | 0 | 7 | 0
Not Completed | 17 | 12 | 1
Not completed — Disease Progression | 7 | 3 | 1
Not completed — Couldn't Start Cycle After Planned Date | 1 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0
Not completed — Other | 4 | 3 | 0
Not completed — Adverse Event | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as a group of participants who received at least 1 dose of the study drug with at least 1 evaluable postbaseline safety data.
Groups:
- PTCL: E7777 9 mcg/kg/Day: Participants with relapsed or refractory PTCL received E7777 9 mcg/kg/day as intravenous infusion, once daily from Day 1 through Day 5 in each treatment cycle until discontinuation or Cycle 8 (each Cycle length = 3 weeks).
- CTCL: E7777 9 mcg/kg/Day: Participants with CTCL received E7777 9 mcg/kg/day as intravenous infusion, once daily from Day 1 through Day 5 in each treatment cycle until discontinuation or Cycle 8 (each Cycle length = 3 weeks).
- Other: E7777 9 mcg/kg/Day: Participant with extranodal NK/T-cell lymphoma received E7777 9 mcg/kg/day as intravenous infusion, once daily from Day 1 through Day 5 in each treatment cycle until discontinuation or Cycle 8 (each Cycle length = 3 weeks).
- Total: Total of all reporting groups
Arm/Group | PTCL: E7777 9 mcg/kg/Day | CTCL: E7777 9 mcg/kg/Day | Other: E7777 9 mcg/kg/Day | Total
Number analyzed (Participants) | 17 | 19 | 1 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (9.16) | 55.3 (15.09) | 70.0 | 60.9 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 1 | 12
  Male | 12 | 13 | 0 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 19 | 1 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 17 | 19 | 1 | 37

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants whose best overall response (BOR) was complete response (CR) or partial response (PR) based on independent review of Efficacy and Safety Evaluation Committee. ORR was assessed according to modified response criteria based on the revised response criteria for malignant lymphoma (Cheson, 2007), skin lesion and peripheral blood disease were assessed according to clinical end points and response criteria in mycosis fungoides and Sezary syndrome (Olsen, 2011). CR: Disappearance of all evidence of disease; PR: Regression of measurable disease and no new sites.
Time Frame: From the date of administration of the first dose of the study drug until completion of the study or treatment discontinuation, up to approximately 3 years 1 month
Population: The full analysis set (FAS) was defined as a group of participants who received at least 1 dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCL: E7777 9 mcg/kg/Day | CTCL: E7777 9 mcg/kg/Day | Other: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 17 | 19 | 0
percentage of participants | 41.2 [18.4 to 67.1] | 31.6 [12.6 to 56.6] |

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS: time between the date of administration of the first dose of the study drug and the date of the first documentation of progressive disease (PD) or death due to any cause (whichever occurred first) based on independent review of Efficacy and Safety Evaluation Committee, assessed by modified response criteria based on the revised response criteria for malignant lymphoma (Cheson, 2007), skin lesion and peripheral blood disease assessed according to clinical end points and response criteria in mycosis fungoides and Sezary syndrome (Olsen, 2011). PD: Any new lesion or unequivocally increase of previously involved sites from nadir. PFS was calculated using Kaplan-Meier method. Participants with no baseline assessments, treatment discontinuation without postbaseline tumor assessments, new anticancer treatment started prior to disease progression, death or PD after more than one missed tumor assessments and participants still on treatment without PD as of data cut-off were censored.
Time Frame: From the date of administration of the first dose of the study drug until date of the first documentation of PD or death due to any cause (whichever occurred first) up to approximately 3 years 1 month
Population: The FAS was defined as a group of participants who received at least 1 dose of the study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PTCL: E7777 9 mcg/kg/Day | CTCL: E7777 9 mcg/kg/Day | Other: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 17 | 19 | 0
months | 2.14 [1.05 to 4.47] | 4.24 [2.56 to NA] — Upper limit of confidence interval could not be estimated due to an insufficient number of events. |

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR: Time between date of first documentation of CR or PR and PD or death due to any cause based on independent review of Efficacy and Safety Evaluation Committee, assessed by modified response criteria based on revised response criteria for malignant lymphoma (Cheson,2007),skin lesion and peripheral blood disease by clinical end points and response criteria in mycosis fungoides and Sezary syndrome(Olsen,2011). DOR was assessed in responders who had CR or PR. CR: Disappearance of all evidence of disease; PR: Regression of measurable disease and no new sites. PD: Any new lesion or unequivocally increase of previously involved sites from nadir. DOR was calculated using Kaplan-Meier method. Participants with new anticancer treatment started prior to disease progression, death or PD after more than one missed tumor assessments and participants still on treatment without PD as of data cut-off were censored.
Time Frame: From the date of first documentation of CR or PR until date of the first documentation of PD or death due to any cause (whichever occurred first) up to approximately 3 years 1 month
Population: The FAS was defined as a group of participants who received at least 1 dose of the study drug. Here "overall number of participants analyzed" signifies responded participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PTCL: E7777 9 mcg/kg/Day | CTCL: E7777 9 mcg/kg/Day | Other: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 7 | 6 | 0
months | 3.09 [0.92 to 4.76] | 4.83 [2.66 to NA] — Upper limit of confidence interval could not be estimated due to an insufficient number of events. |

4. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as time between the date of administration of the first dose of the study drug and the date of first documentation PR or CR based on independent review of Efficacy and Safety Evaluation Committee. PR or CR were assessed according to modified response criteria based on the revised response criteria for malignant lymphoma (Cheson, 2007), skin lesion and peripheral blood disease were assessed according to clinical end points and response criteria in mycosis fungoides and Sezary syndrome (Olsen, 2011). TTR was only conducted among responders who had experienced CR or PR. CR: Disappearance of all evidence of disease; PR: Regression of measurable disease and no new sites.
Time Frame: From the date of administration of the first dose of the study drug until date of the first documentation of PR or CR or death due to any cause (whichever occurred first) up to approximately 3 years 1 month
Population: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | PTCL: E7777 9 mcg/kg/Day | CTCL: E7777 9 mcg/kg/Day | Other: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 7 | 6 | 0
months | 1.28 [1.0 to 2.1] | 2.12 [1.0 to 4.6] |

5. Secondary Outcome: CR Rate
Description: CR rate was defined as the percentage of participants whose BOR was CR based on independent review of Efficacy and Safety Evaluation Committee. CR was assessed according to modified response criteria based on the revised response criteria for malignant lymphoma (Cheson, 2007), skin lesion and peripheral blood disease were assessed according to clinical end points and response criteria in mycosis fungoides and Sezary syndrome (Olsen, 2011). CR: Disappearance of all evidence of disease.
Time Frame: as for outcome 1
Population: The FAS was defined as a group of participants who received at least 1 dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCL: E7777 9 mcg/kg/Day | CTCL: E7777 9 mcg/kg/Day | Other: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 17 | 19 | 0
percentage of participants | 5.9 [0.1 to 28.7] | 0 [0.0 to 17.6] |

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the date of administration of the first dose of the study drug and the date of death due to any cause. Participants who were alive at cut-off were censored.
Time Frame: From date of administration of the first dose of the study drug until the date of death due to any cause up to approximately 3 years 1 month
Population: The FAS was defined as a group of participants who received at least 1 dose of the study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PTCL: E7777 9 mcg/kg/Day | CTCL: E7777 9 mcg/kg/Day | Other: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 17 | 19 | 0
months | 11.79 [4.11 to 19.29] | 31.87 [16.85 to NA] — Upper limit of confidence interval could not be estimated due to an insufficient number of events. |

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From the date of administration of the first dose of the study drug up to 30 days after the last dose of study drug (approximately up to 3 years 1 month)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PTCL: E7777 9 mcg/kg/Day | CTCL: E7777 9 mcg/kg/Day | Other: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 17 | 19 | 1
Participants
  TEAEs | 17 | 19 | 1
  SAEs | 9 | 8 | 0

8. Secondary Outcome: Cmax: Maximum Observed Serum Concentration for E7777
Time Frame: Cycle 1 Day 1: 0-240 minutes post-infusion; Cycle 3 and 5 Day 1: 0-120 minutes post-infusion (each Cycle length = 3 weeks)
Population: The pharmacokinetic (PK) analysis set was defined as a group of participants who received at least 1 dose of the study drug with at least 1 serum concentration data, and included participants who had been taken frequent blood sampling for non-compartment analysis. PK-evaluable population where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- PTCL and CTCL Participants: E7777 9 mcg/kg/Day: Participants with relapsed or refractory PTCL and CTCL received E7777 9 mcg/kg/day as intravenous infusion, once daily from Day 1 through Day 5 in each treatment cycle until discontinuation or Cycle 8 (each Cycle length = 3 weeks).
Arm/Group | PTCL and CTCL Participants: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 11
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 132 (43.1)
  Cycle 3 Day 1: number analyzed (Participants) | 1
  Cycle 3 Day 1 | 142 (NA) — Standard deviation could not be calculated because only one participant was analysed.
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 140 (NA) — Standard deviation could not be calculated because only one participant was analysed.

9. Secondary Outcome: Tmax: Time to Reach the Cmax for E7777
Time Frame: as for outcome 8
Population: The PK analysis set was defined as a group of participants who received at least 1 dose of the study drug with at least 1 serum concentration data, and included participants who had been taken frequent blood sampling for non-compartment analysis. PK-evaluable population where data at specified time points was available.
Measure: Median (Full Range); unit: minutes
Arm/Group | PTCL and CTCL Participants: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 11
minutes
  Cycle 1 Day 1 | 63.00 [59.00 to 99.00]
  Cycle 3 Day 1: number analyzed (Participants) | 1
  Cycle 3 Day 1 | 65.00 [NA to NA] — Full range could not be calculated because only one participant was analysed.
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 80.00 [NA to NA] — Full range could not be calculated because only one participant was analysed.

10. Secondary Outcome: AUC(0-t ): Area Under the Serum Concentration-time Curve From Time 0 to the Last Measurable Point for E7777
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nanogram*minute permilliliter(ng*min/mL)
Arm/Group | PTCL and CTCL Participants: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 11
nanogram*minute permilliliter(ng*min/mL)
  Cycle 1 Day 1 | 17600 (8040)
  Cycle 3 Day 1: number analyzed (Participants) | 1
  Cycle 3 Day 1 | 15800 (NA) — Standard deviation could not be calculated because only one participant was analysed.
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 16500 (NA) — Standard deviation could not be calculated because only one participant was analysed.

11. Secondary Outcome: AUC(0-inf): Area Under the Serum Concentration-time Curve From Time 0 to Infinity for E7777
Description: 11 participants were included in the PK analysis, however AUC(0-inf), could not be estimated for 1 participant due to insufficient data for elimination rate constant.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*min/m
Arm/Group | PTCL and CTCL Participants: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 11
ng*min/m
  Cycle 1 Day 1: number analyzed (Participants) | 10
  Cycle 1 Day 1 | 23000 (7830)
  Cycle 3 Day 1: number analyzed (Participants) | 0
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 21400 (NA) — Standard deviation could not be calculated because only one participant was analysed.

12. Secondary Outcome: Mean Residence Time (MRT) for E7777
Description: 11 participants were included in the PK analysis, however MRT, could not be estimated for 1 participant due to insufficient data for elimination rate constant.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PTCL and CTCL Participants: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 11
minutes
  Cycle 1 Day 1: number analyzed (Participants) | 10
  Cycle 1 Day 1 | 136 (29.2)
  Cycle 3 Day 1: number analyzed (Participants) | 0
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 105 (NA) — Standard deviation could not be calculated because only one participant was analysed.

13. Secondary Outcome: t1/2: Terminal Elimination Phase Half-life for E7777
Description: 11 participants were included in the PK analysis, however t1/2, could not be estimated for 1 participant due to insufficient data for elimination rate constant.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PTCL and CTCL Participants: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 11
minutes
  Cycle 1 Day 1: number analyzed (Participants) | 10
  Cycle 1 Day 1 | 96.0 (19.6)
  Cycle 3 Day 1: number analyzed (Participants) | 1
  Cycle 3 Day 1 | 116 (NA) — Standard deviation could not be calculated because only one participant was analysed.
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 69.2 (NA) — Standard deviation could not be calculated because only one participant was analysed.

14. Secondary Outcome: CL: Total Clearance for E7777
Description: 11 participants were included in the PK analysis, however CL, could not be estimated for 1 participant due to insufficient data for elimination rate constant.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliter per minute per kilogram
Arm/Group | PTCL and CTCL Participants: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 11
milliter per minute per kilogram
  Cycle 1 Day 1: number analyzed (Participants) | 10
  Cycle 1 Day 1 | 0.465 (0.250)
  Cycle 3 Day 1: number analyzed (Participants) | 0
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 0.421 (NA) — Standard deviation could not be calculated because only one participant was analysed.

15. Secondary Outcome: Vz: Volume of Distribution at Terminal Phase for E7777
Description: 11 participants were included in the PK analysis, however Vz, could not be estimated for 1 participant due to insufficient data for elimination rate constant.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliliter per kilogram (mL/kg)
Arm/Group | PTCL and CTCL Participants: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 11
milliliter per kilogram (mL/kg)
  Cycle 1 Day 1: number analyzed (Participants) | 10
  Cycle 1 Day 1 | 59.0 (17.4)
  Cycle 3 Day 1: number analyzed (Participants) | 0
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 42.0 (NA) — Standard deviation could not be calculated because only one participant was analysed.

16. Secondary Outcome: Vss: Volume of Distribution at Steady State for E7777
Description: 11 participants were included in the PK analysis, however Vss, could not be estimated for 1 participant due to insufficient data for elimination rate constant.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | PTCL and CTCL Participants: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 11
mL/kg
  Cycle 1 Day 1: number analyzed (Participants) | 10
  Cycle 1 Day 1 | 57.4 (13.5)
  Cycle 3 Day 1: number analyzed (Participants) | 0
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 44.1 (NA) — Standard deviation could not be calculated because only one participant was analysed.

17. Secondary Outcome: Rac (Cmax): Accumulation Ratio of Cmax for E7777
Description: Accumulation Ratio of Cmax was calculated as RAC (Cmax) on Cycle 3 Day 1 divided by RAC (Cmax) on Cycle 1 Day 1, and RAC (Cmax) on Cycle 5 Day 1 divided by RAC (Cmax) on Cycle 1 Day 1.
Time Frame: as for outcome 8
Population: PK analysis set: group of participants who received at least 1 dose of study drug with at least 1 serum concentration data, and included participants who had taken frequent blood sampling for non-compartment analysis. Overall number of participants analyzed is number of participants with evaluable data at Cycle 1 Day 1 and at Cycles 3 and 5 Day 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PTCL and CTCL Participants: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 1
ratio
  Cycle 3 Day 1 | 0.993 (NA) — Standard deviation could not be calculated because only one participant was analysed.
  Cycle 5 Day 1 | 0.979 (NA) — Standard deviation could not be calculated because only one participant was analysed.

18. Secondary Outcome: Rac (AUC): Accumulation Ratio of AUC for E7777
Description: Accumulation ratio of AUC was calculated as RAC (AUC) on Cycle 3 Day 1 divided by RAC (AUC) on Cycle 1 Day 1, and RAC (AUC) on Cycle 5 Day 1 divided by RAC (AUC) on Cycle 1 Day 1.
Time Frame: as for outcome 8
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PTCL and CTCL Participants: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 1
ratio
  Cycle 3 Day 1: number analyzed (Participants) | 0
  Cycle 5 Day 1 | 0.827 (NA) — Standard deviation could not be calculated because only one participant was analysed.

19. Secondary Outcome: Number of Participants With Positive Anti-E7777 and Anti-IL-2 Antibodies
Time Frame: Cycles 1, 2, 3, 5, 8: Day 1 pre-dose; at treatment discontinuation or completion (Cycle 8 Day 21) (each Cycle length = 3 weeks)
Population: The pharmacodynamics (PD) analysis set was defined as a group of participants who received at least 1 dose of the study drug with at least 1 each of evaluable pre- and post-baseline PD data. Participants who were evaluable for this measure at given time point were included for the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | PTCL: E7777 9 mcg/kg/Day | CTCL: E7777 9 mcg/kg/Day | Other: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 17 | 19 | 1
Participants
  Anti-E7777 antibody: Cycle 1 Day 1 | 11 | 13 | 1
  Anti-E7777 antibody: Cycle 2 Day 1: number analyzed (Participants) | 11 | 14 | 1
  Anti-E7777 antibody: Cycle 2 Day 1 | 5 | 11 | 0
  Anti-E7777 antibody: Cycle 3 Day 1: number analyzed (Participants) | 8 | 13 | 0
  Anti-E7777 antibody: Cycle 3 Day 1 | 3 | 11 |
  Anti-E7777 antibody: Cycle 5 Day 1: number analyzed (Participants) | 4 | 11 | 0
  Anti-E7777 antibody: Cycle 5 Day 1 | 1 | 10 |
  Anti-E7777 antibody: Cycle 8 Day 1: number analyzed (Participants) | 0 | 7 | 0
  Anti-E7777 antibody: Cycle 8 Day 1 |  | 7 |
  Anti-E7777 antibody: Discontinuation/Completion: number analyzed (Participants) | 16 | 18 | 1
  Anti-E7777 antibody: Discontinuation/Completion | 10 | 15 | 1
  Anti-IL-2 antibody: Cycle 1 Day 1 | 1 | 1 | 0
  Anti-IL-2 antibody: Cycle 2 Day 1: number analyzed (Participants) | 11 | 14 | 1
  Anti-IL-2 antibody: Cycle 2 Day 1 | 2 | 4 | 0
  Anti-IL-2 antibody: Cycle 3 Day 1: number analyzed (Participants) | 8 | 13 | 0
  Anti-IL-2 antibody: Cycle 3 Day 1 | 2 | 11 |
  Anti-IL-2 antibody: Cycle 5 Day 1: number analyzed (Participants) | 4 | 11 | 0
  Anti-IL-2 antibody: Cycle 5 Day 1 | 1 | 10 |
  Anti-IL-2 antibody: Cycle 8 Day 1: number analyzed (Participants) | 0 | 7 | 0
  Anti-IL-2 antibody: Cycle 8 Day 1 |  | 7 |
  Anti-IL-2 antibody: Discontinuation/Completion: number analyzed (Participants) | 16 | 18 | 1
  Anti-IL-2 antibody: Discontinuation/Completion | 3 | 15 | 0

20. Secondary Outcome: Number of Participants With Positive Neutralizing Activity of Anti-E7777 Antibody
Time Frame: as for outcome 19
Population: The PD analysis set was defined as a group of participants who received at least 1 dose of the study drug with at least 1 each of evaluable pre- and post-baseline PD data. Participants who were evaluable for this measure at given time point were included for the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | PTCL: E7777 9 mcg/kg/Day | CTCL: E7777 9 mcg/kg/Day | Other: E7777 9 mcg/kg/Day
Number analyzed (Participants) | 17 | 19 | 1
Participants
  Cycle 1 Day 1 | 0 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 11 | 14 | 1
  Cycle 2 Day 1 | 2 | 9 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 8 | 13 | 0
  Cycle 3 Day 1 | 2 | 11 |
  Cycle 5 Day 1: number analyzed (Participants) | 4 | 11 | 0
  Cycle 5 Day 1 | 1 | 8 |
  Cycle 8 Day 1: number analyzed (Participants) | 0 | 7 | 0
  Cycle 8 Day 1 |  | 6 |
  Discontinuation/Completion: number analyzed (Participants) | 16 | 18 | 1
  Discontinuation/Completion | 8 | 12 | 0

ADVERSE EVENTS:
Time Frame: From the date of administration of the first dose of the study drug up to 30 days after the last dose of study drug (approximately up to 3 years 1 month)
Arm/Group | PTCL: E7777 9 mcg/kg/Day | CTCL: E7777 9 mcg/kg/Day | Other: E7777 9 mcg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/17 | 1/19 | 0/1
Serious Adverse Events (participants affected / at risk) | 9/17 | 8/19 | 0/1
Other Adverse Events (participants affected / at risk) | 17/17 | 19/19 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTCL: E7777 9 mcg/kg/Day (N=17) | CTCL: E7777 9 mcg/kg/Day (N=19) | Other: E7777 9 mcg/kg/Day (N=1)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 4 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTCL: E7777 9 mcg/kg/Day (N=17) | CTCL: E7777 9 mcg/kg/Day (N=19) | Other: E7777 9 mcg/kg/Day (N=1)
Lymphopenia (Blood and lymphatic system disorders) | 14 | 11 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0
Disorder of orbit (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Eczema eyelids (Eye disorders) | 1 | 0 | 0
Photopsia (Eye disorders) | 0 | 1 | 0
Retinal exudates (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 10 | 0
Nausea (Gastrointestinal disorders) | 5 | 6 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Perianal erythema (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 9 | 7 | 1
Malaise (General disorders) | 4 | 8 | 0
Oedema peripheral (General disorders) | 5 | 3 | 0
Fatigue (General disorders) | 3 | 1 | 0
Generalised oedema (General disorders) | 0 | 3 | 0
Face oedema (General disorders) | 1 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Puncture site pain (General disorders) | 0 | 1 | 0
Vessel puncture site erythema (General disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Angular cheilitis (Infections and infestations) | 1 | 1 | 0
Lung infection (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Genital candidiasis (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Skin candida (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 13 | 15 | 1
Alanine aminotransferase increased (Investigations) | 13 | 15 | 0
Gamma-glutamyltransferase increased (Investigations) | 9 | 7 | 1
Lipase increased (Investigations) | 6 | 4 | 0
Weight increased (Investigations) | 4 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 3 | 1
Amylase increased (Investigations) | 3 | 2 | 0
Blood cholesterol increased (Investigations) | 3 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 3 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood fibrinogen decreased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 1 | 0 | 0
Cytomegalovirus test positive (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 | 14 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 5 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 5 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 4 | 0
Delirium (Psychiatric disorders) | 1 | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Prostatic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 4 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 3 | 0
Hot flush (Vascular disorders) | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT02676778/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT02676778/SAP_001.pdf